CLINICAL TRIAL: NCT01877798
Title: Venoarterial PCO2 Difference /Arteriovenous O2 Content Difference Ratio as Goal of Early Severe Sepsis and Septic Shock Therapy
Brief Title: Venoarterial PCO2 Difference /Arteriovenous O2 Content Difference Ratio as Goal of Early Septic Shock Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCSS
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- △PCO2/Ca-vO2 (Experimental): △PCO2/Ca-vO2 directed group
  Interventions: Procedure: volume resuscitation, vasoactive drug
- ScvO2 (Experimental): ScvO2 directed group
  Interventions: Procedure: volume resuscitation, vasoactive drug

INTERVENTIONS:
Procedure: volume resuscitation, vasoactive drug

SUMMARY:
Reducing tissue hypoxia is the ultimate goal of severe sepsis and septic shock therapy.Venoarterial PCO2 difference /arteriovenous O2 content difference ratio (△PCO2/Ca-vO2) is considered to be a good indicator of global anaerobic metabolism.The purpose of this study was to compare the efficacy of △PCO2/Ca-vO2 and central venous oxygen saturation (ScvO2) in the treatment of severe sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

* severe sepsis and septic shock patients

Exclusion Criteria:

* <18 years old
* pregnant and breast-feed woman
* AMI
* cerebral hemorrhage
* contraindication for central venous catheter or arterial catheter;
* brainstem death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital critical care medicine, Beijing, China

REFERENCES:
- [Derived] Su L, Tang B, Liu Y, Zhou G, Guo Q, He W, Wang C, Zhuang H, Jiang L, Qin L, Deng Q, Shuai W, Zhang L, Wang X, Su J, Ma S, Liu D, Long Y. P(v-a)CO2/C(a-v)O2-directed resuscitation does not improve prognosis compared with SvO2 in severe sepsis and septic shock: A prospective multicenter randomized controlled clinical study. J Crit Care. 2018 Dec;48:314-320. doi: 10.1016/j.jcrc.2018.09.009. Epub 2018 Sep 11. PMID 30278407